CLINICAL TRIAL: NCT01586325
Title: A Phase Ib, Randomized, Double-Blind, Placebo-Controlled Trial in Asian Genotype 1 Chronic HCV-Infected Subjects to Determine the Safety, Tolerability, Pharmacokinetics and Antiviral Activity of Repeated Doses of JNJ-47910382 Given in Different Doses and Dose Regimens
Brief Title: A Study of the Safety, Tolerability, Pharmacokinetics, and Antiviral Activity of JNJ-47910382 at Different Doses and Dose Regimens in Asian Genotype-1, Chronic, HCV-Infected Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Because of many competing trials using the same mechanism of action, but being further advanced in development
Sponsor: Janssen R&D Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR100718; 47910382HPC1003 (Other: Janssen R&D Ireland)
Record Dates: First submitted 2012-04-24; First posted 2012-04-26 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Chronic Hepatitis C Infection
Keywords: Chronic hepatitis C infection; Asian genotype 1 chronic hepatitis C infection; JNJ-47910382; Non-structural protein 5A (NS5A) inhibitor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Panel 1 (Experimental): Study participants will receive double-blind treatment with JNJ-47910382 30 mg or matching placebo. Participants in each of Panel will be treated sequentially (ie, participants in Panel 1 will be treated before participants in Panel 2, participants in Panel 2 will be treated before participants in Panel 3).
  Interventions: Drug: JNJ-47910382 30 mg; Drug: Placebo
- Panel 2 (Experimental): Study participants will receive double-blind treatment with JNJ-47910382 90 mg or matching placebo. Participants in each of Panel will be treated sequentially.
  Interventions: Drug: JNJ-47910382 90 mg; Drug: Placebo
- Panel 3 (Experimental): Study participants will receive double-blind treatment with JNJ-47910382 200 mg (maxiumum dose) or matching placebo. Participants in each of Panel will be treated sequentially.
  Interventions: Drug: JNJ-47910382 200 mg; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-47910382 30 mg — JNJ-47910382 30 mg (0.6 mL of an oral suspension of 50 mg/mL of JNJ-47910382) administered once daily as monotherapy for 5 days.
  Arms: Panel 1
Drug: JNJ-47910382 90 mg — JNJ-47910382 90 mg (1.8 mL of an oral suspension of 50 mg/mL of JNJ-47910382) administered once daily as monotherapy for 5 days.
  Arms: Panel 2
Drug: JNJ-47910382 200 mg — JNJ-47910382 200 mg (4 mL of an oral suspension of 50 mg/mL of JNJ-47910382) administered once daily as monotherapy for 5 days.
  Arms: Panel 3
Drug: Placebo — Matching Placebo administered once daily as monotherapy for 5 days.

SUMMARY:
The purpose of this study is to determine the safety, tolerability, pharmacokinetics (how a drug is absorbed and distributed in the body), and intrinsic antiviral activity of JNJ-47910382 after 5 consecutive days of administration in chronic, hepatitis C virus (HCV)-genotype-1-infected patients at different doses and dose regimens.

DETAILED DESCRIPTION:
This is a double-blind (neither physician nor patient knows the name of the assigned drug), randomized (patients are assigned by chance to treatment groups) placebo-controlled study. A placebo is an inactive substance that is compared with a drug to test whether the drug has a real effect. The study population will consist of Asian treatment-naive genotype-1, chronic HCV-infected patients. The trial will involve a screening period at a maximum of 6 weeks before baseline, a 9-day treatment period (with 5 days of actual medication intake) and a 4-week follow-up period. Patients will be divided into 3 panels of 8 patients (Panel 1) or 5 patients (Panels 2 and 3). Treatment will be initiated in each panel of patients sequentially. In each panel, patients will receive JNJ-47910382 or placebo during 5 consecutive days. JNJ-47910382, or placebo, will be administered once daily. Treatments will be taken by mouth and with standardized meals in all dosing regimens. Patient safety will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Documented chronic HCV infection (diagnosis of hepatitis C >= 6 months before the screening period)
* HCV geno- and subtype of 1a or 1b (Panel 1) or 1b (Panels 2 and 3)
* Patient has never received pegylated interferon, ribavirin, or any other approved or investigational antiviral treatment for chronic HCV infection
* Patient with HCV ribonucleic acid (RNA) level of >100,000 IU/mL at screening (as assessed by standard quantitative in vitro nucleic acid amplification assay)
* A Body Mass Index (BMI, weight in kg divided by the square of height in meters) of 18.0 to 32.0 kg/m2, extremes included
* A body weight above 50 kg
* Normal 12-lead electrocardiogram (ECG) at screening

Exclusion Criteria:

* Evidence of or documented liver cirrhosis
* Evidence of decompensated liver disease
* Evidence of any other cause of significant liver disease in addition to hepatitis C
* History or evidence of current use of alcohol, barbiturate, amphetamine, recreational or narcotic drug use, which in the Investigator's opinion would compromise patient's safety and/or compliance with the study procedures
* A positive urine drug (with exclusion of methadone or equivalent) test at study screening
* Patient with protocol-defined laboratory abnormalities at screening
* Patient coinfected with HIV-1 or HIV-2, or hepatitis A or B virus infection, or active tuberculosis at study screening
* Patient infected/coinfected with non-genotype 1 HCV at study screening
* Patient with any cardiac disease at screening, or any active clinically significant disease (eg, cardiac dysfunction, cardio(myo)pathy, cardiac insufficiency), or medical history or physical examination findings during screening that, in the Investigator's opinion, would compromise the outcome of the trial
* Patient having uncontrolled/unstable disease such as diabetes, epilepsy, a manifest psychiatric disease, or thyroid disease or disorders
* Patient with non-stable methadone (or equivalent drug) use

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-05-25 (Actual); Primary Completion 2014-04-21 (Actual); Study Completion 2014-04-21 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HCV RNA levels over time during the 5-day treatment regimen | Up to 4 weeks after the last dose of study medication.
Number of participants with HCV RNA levels below the limit of detection | Up to 4 weeks after the last dose of study medication.

SECONDARY OUTCOMES:
Mean plasma concentrations of JNJ-47910382 | Up to Day 9 of each treatment period.
Maximum observed plasma concentration of JNJ-47910382 | Up to Day 9 of each treatment period.
Minimum observed plasma concentration of JNJ-47910382 | Up to Day 9 of each treatment period
Time to reach the maximum plasma concentration of JNJ-47910382 | Up to Day 9 of each treatment period.
Area under the plasma concentration-time curve from time 0 to 24 hours of JNJ-47910382 | Up to Day 9 of each treatment period.
Average steady-state plasma concentration of JNJ-47910382 | Up to Day 9 of each treatment period.
Terminal elimination half life of JNJ-47910382 | Up to Day 9 of each treatment period.
The number of participants affected by an adverse event | Up to 30 days after the last dose of study medication

CONTACTS AND LOCATIONS:
Overall Officials: Janssen R&D Ireland Clinical Trial, Study Director — Janssen R&D Ireland
Locations (5):
- Taiwan (5):
  - Kaohsiung City
  - Niaosung, Kaohsiung
  - Taichung
  - Tainan
  - Taipei